CLINICAL TRIAL: NCT04220944
Title: Microwave Ablation Combined With Simultaneous TACE Plus Sintilimab for Unresectable HCC.
Brief Title: Combined Locoregional Treatment With Immunotherapy for Unresectable HCC.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR-2019B
Record Dates: First submitted 2019-12-29; First posted 2020-01-07 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Carcinoma
Keywords: HCC; Microwave ablation; TACE; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Locoregional therapies combined with Anti-PD-1 antibody (Experimental): Percutaneous microwave ablation combined with simultaneous TACE was performed. Sintilimab will be initiated on day 3-7 after the first locoregional therapies. Sintilimab will be administered every three weeks (200mg fixed dose IV) until disease progression for up to one year.The second locoregional procedure will be repeated according to the enhanced CT images.
  Interventions: Drug: Sintilimab; Procedure: Microwave Ablation; Procedure: TACE

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (200mg) was administered intravenously over 30-60 min every 3 weeks.
  Other Names: Sintilimab injection, 308004
Procedure: Microwave Ablation — The ablation area should covered at least two thirds the size of the nodules.
Procedure: TACE — Patient was treated with epirubicin lipiodol emulsion(Epirubicin 40mg, Lipiodol 10ml).Embolic materials such as gelfoam or microsphere was aslo administered until complete stasis in segmental or subsegmental arterial branches.

SUMMARY:
Efficacy and Safety of Locoregional treatments Combined With PD-1 Inhibitor in Patients With Unresectable Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is the most frequent primary and ranked as the sixth most common neoplasm and the third leading cause of cancer death.

Percutaneous ablation and TACE are the effective locoregional treatments for the patient with HCC. Moreover, some studies suggested that TACE combined with ablation could further improve the survival rate and reduce the post-operation complication.

Although PD-1 inhibitor was approved by FDA for HCC, the latest RCT indicated that no significant difference was found in the ORR and PFS between the groups of PD-1 inhibitor and Sorafenib.

Therefore, this study aims to assess the efficacy and safety of microwave ablation combined with simultaneous TACE plus PD-1 inhibitor for the non-resectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 80 years old and life expectancy of at least 12 weeks.;
2. Clinically or histologically diagnosed as HCC and the diameter of target tumor lesion ≥ 5 cm;
3. Child-pugh classification A or B (score < 7);
4. BCLC Staging as B or C;
5. ECOG 0-1;
6. Patients voluntarily entered the study and signed informed consent form (ICF).

Exclusion Criteria:

1. History of treatment with any local treatment (exception of liver transplantation), systemic .anti-cancer therapy, or immunotherapy;
2. The surgeon assessed that the tumor lesion was not unsuitable for microwave ablation;
3. Any contraindications for hepatic embolization procedures:

   1. Known hepatofugal blood flow;
   2. Total thrombosis of main portal vein.
4. The tumor thrombus of main portal vein, IVC or right atrium;
5. Tumor burden ≥ 70% of liver volume; and no measurable site of disease as defined by modified RECIST (mRECIST) criteria with spiral CT scan or MRI;
6. Subjects with chronic HBV infection have HBV DNA viral load > 100 IU/mL at screening, and have not received antiviral therapy prior to initiation of study therapy; In addition, coinfection of HBV and HCV;
7. The alcoholic or pregnant women;
8. Patients with second primary cancer or history of other cancer within 3 years;
9. Diagnosis of active autoimmune disease, immunodeficiency, or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Sintilimab-monotherapy treatment;
10. Blood count, liver function: Haemoglobin < 9.0 g/dL, white cell count < 1.0 x10^9/L; Total bilirubin > 3 mg/dL; Aspartate Aminotransferase (SGOT) or Alanine aminotransferase (SGPT) > 5 x upper normal limit (ULN), Albumin < 2.8g/dL; International normalized ratio (INR) >2.3;
11. Renal function dysfunction: Serum Creatinine >2 mg/dL or creatinine clearance (CrCl) < 30 mL/min (if using the Cockcroft-Gault formula ); and severe heart, lung, brain or other organ disease;
12. Non-compliance with TACE or ablation procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Observation period max 18 months
  Progression according to mRECIST for HCC.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | max 18 months
  Objective Response Rate according to mRECIST for HCC
Time to Progression (TTP) | max 18 months
  It is defined as the time from first locoregional therapy to the date of the first documented tumor progression according to the definition above.
Overall survival (OS) | max 18 months
  Overall survival is defined as the time from first locoregional therapy until death
Incidence of Treatment Emergent Adverse Events as assessed by NCI CTCAE V5.0 (Safety and Tolerability) | max 18 months
  Data will be obtained on vital signs, clinical parameters and feasibility of the regimen

CONTACTS AND LOCATIONS:
Overall Officials: zhiping Yan, MD, Study Director — Department of Interventional Radiology, Zhongshan Hospital, Fudan University
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No